CLINICAL TRIAL: NCT03165370
Title: The Study of the Relationship of Insomnia in the Traditional Chinese Medicine and Western Medicine at Local Clinic
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Ching-Liang Hsieh, Attending Physician, China Medical University Hospital
Other Study IDs: CRREC-106-028
Record Dates: First submitted 2017-05-18; First posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Insomnia: those with unsatisfactory sleep quantity and/or quality (difficulty with sleep induction, awakenings during the night, early morning awakening, total sleep time, and overall quality of sleep), complaint of a minimum frequency (at least three times a week) and duration (1 month), marked distress caused by the sleep problem and/or interference with ordinary activities of daily living

SUMMARY:
Insomnia is one of the most main diseases of civilization in the world, which chronic insomnia is up to 30% in Taiwan under the latest statistics and a common disease which appears to sleep difficultly, sleep interrupted, wake up early or wake up still tired. Long-term persistence of these symptoms will lead to the occurrence of mental illness and then affect people's emotional behavior and cognitive memory, showing that insomnia is an important modern health issues. Recently, "individual response patterns" was proposed by modern medicine. This thinking process and spirit seems to be compatible with the traditional Chinese medicine (TCM) therapy of "Differential Treatment". The purpose of this study, the Athens Insomnia Scale (AIS), commonly used to quickly screen for insomnia patients and the evaluation of Western medicine efficacy in Western medicine clinic, and investigation of Syndrome Type of TCM to find out whether with Syndrome Type of TCM and AIS in the associated factors, and confirm the necessity and importance of Syndrome Type of TCM, for future reference and basis for the development of integrated medicine.

In the cross-section study with an interview on survey, sampling Miaoli County an Chinese medicine clinic, in line with standard sampling of 200 patients with insomnia were recruited. The questionnaires contained two instruments including Athens Insomnia Scale (AIS), and Syndrome Type of TCM questionnaire. Cross-table, chi-square test, variance analysis and Pearson product-moment correlation was used to find the relation.

DETAILED DESCRIPTION:
Insomnia is a common sleep disturbance, there were more than a quarter of people with sleep disorders, the prevalence with more and higher, seriously affecting the health and quality of life. The Athens Insomnia Scale (referred to as AIS) can help physicians more accurately diagnose and understand the state of insomnia patients. The purpose of this study was investigated the correlation among the disease status, treatment and AIS assessment, hoping enough traditional Chinese physician and Western physician's clinical reference. Methods: This study used the cross-sectional questionnaire survey with the convenience sampling method. Screened 200 patients according to the diagnostic criteria for insomnia and conducted a survey from the local clinic at Miaoli County.

ELIGIBILITY:
Inclusion Criteria:

* Compliance with the International Statistical Classification of Diseases and Related Health Problems (ICD)-10 and the Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV and other international standards in the diagnosis of non-organic insomnia criteria to determine the main diagnosis and secondary diagnosis of insomnia: A. Complaint of difficulty initiating sleep, difficulty maintaining sleep, or waking up too early, or sleep that is chronically nonrestorative or poor in quality. B. Any sleep difficulty at least three times a week and during the period of the last month. C. Over concerns or worries about sleep. D. The night time sleep difficulty is related to daytime impairment: mood disturbance or social and vocational dysfunction
* Cooperation with physician voluntarily, communication with physician normally

Exclusion Criteria:

* Teenagers and babies
* Insomnia associated with other sleep disorders most commonly includes sleep related breathing disorders (e.g.,obstructive sleep apnea), movement disorders (e.g.,restless legs or periodic limb movements during sleep) or circadian rhythm sleep disorders;
* Insomnia due to medical or psychiatric disorders (Schizophrenia, paranoia, affective psychosis, bipolar disorder, depression, organic psychosis like brain injury, epilepsy, dementia and so on), or to drug/substance (comorbid insomnia); and
* Primary insomnias including psychophysiological, idiopathic, and paradoxical insomnias.
* Lack of intelligence or other reasons it is difficult to correctly fill the questionnaire

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: an Chinese medicine clinic at Miaoli County
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-05-19 (Actual); Primary Completion 2018-05-04 (Estimated); Study Completion 2018-05-04 (Estimated)

PRIMARY OUTCOMES:
Questionnaires and Data analysis | Patients were estimated any sleep difficulty during the period of last 4 weeks and then finished record about 15-20 minutes. A copy was done after 2 weeks. From date of randomization until the date of final documented progression, assessed 2 months.
  Scores for each sleep dimension on the AIS questionnaire compared to Syndrome Type of TCM questionnaire. The AIS questionnaire contains 8 items which are rated on 0-3 scale ("0" means "no problem", "1" means "mild problem", "2" means "marked problem", "3" means "severe problem"). For each dimension, item scores are coded, summed, and transformed on to a scale from 0 (best sleep) to 24 (worst sleep) as an individual's sleep outcome. Syndrome Type of TCM questionnaire contains 6 patterns: pattern of yin deficiency with effulgent fire, pattern of deficiency of both heart and spleen, pattern of liver depression transforming into fire, pattern of phlegm-heat harassing internally, pattern of heart and gallbladder qi insufficiency, the other patterns as well and case numbers are counted as an TCM pattern's outcome. Finally, study the distribution law of insomnia's TCM pattern identification and relative factors of AIS.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Liang Hsieh, Principal Investigator — China Medical University Hospital
Locations (1):
- Zhunan Ho-Te Chinese medicine clinic, Miaoli County, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chiu HY, Chang LY, Hsieh YJ, Tsai PS. A meta-analysis of diagnostic accuracy of three screening tools for insomnia. J Psychosom Res. 2016 Aug;87:85-92. doi: 10.1016/j.jpsychores.2016.06.010. Epub 2016 Jun 25. PMID 27411756